CLINICAL TRIAL: NCT02796989
Title: The Impact of Modified Wheat Bran on Carbohydrate Fermentation in the Colon in Healthy and Obese Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: s58346
Record Dates: First submitted 2016-05-27; First posted 2016-06-13 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy; Obese
MeSH Terms: conditions — Obesity | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy - Wheat Bran (Active Comparator): Wheat bran 20 g each day
  Interventions: Dietary Supplement: Wheat bran
- Healthy - Placebo (Placebo Comparator): Placebo 20 g each day
  Interventions: Dietary Supplement: Placebo
- Obese - Wheat bran (Active Comparator): Wheat bran 20 g each day
  Interventions: Dietary Supplement: Wheat bran
- Obese - Placebo (Placebo Comparator): Placebo 20 g each day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wheat bran — 20 g each day
  Arms: Healthy - Wheat Bran; Obese - Wheat bran
Dietary Supplement: Placebo — 20 g each day
  Arms: Healthy - Placebo; Obese - Placebo

SUMMARY:
During this project the effect of modified wheat bran on colon health and systemic health will be evaluated in a long-term intervention study in healthy and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* BMI between 18 and 25 kg/m² OR higher than 30 kg/m²
* Regular diet
* Not dieting

Exclusion Criteria:

* Use of antibiotics in the month preceding the study
* Diabetes Type 1 or 2
* Abdominal surgery (except from appendectomy)
* Use of medication that affects the gastrointestinal tract during the last 2 weeks prior to the study including spasmolytics, anti-diarrhoea medication, anti-constipation medication
* Use of pre- or probiotic supplements in the month preceding the study
* Chronic gastrointestinal diseases, such as inflammatory bowel disease (Crohn's disease, ulcerative colitis), irritable bowel disease…
* Pregnancy or lactation
* Blood donation in the last 3 months
* Abnormal Hb-level (Standard range between 14 and 18 g/dL for men and between 12 and 16 g/dL for women)
* Participation in clinical studies involving radiation exposure in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The incremental plasma short-chain fatty acid concentrations will be measured using GC-FID after an intervention with wheat bran/placebo | 1 month

SECONDARY OUTCOMES:
Changes in glucose levels (mg/dL) | 1 month
Changes in insulin levels (pmol/L) | 1 month
Changes in cholesterol levels (mg/dL) | 1 month
Changes in free fatty acids levels (mmol/L) | 1 month
Changes in triglyceride levels (mg/dL) | 1 month
Gut permeability using 51-Cr-EDTA | 1 month
Total gastrointestinal transit time | 1 month
Changes in gut microbiota before and after the intervention using 16S rRNA sequencing | 1 month
Changes in metabolite patterns in the feces before and after the intervention using gas chromatography coupled to mass spectrometry | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium